CLINICAL TRIAL: NCT06388642
Title: A Study to Evaluate the Pharmacokinetics of Afamelanotide in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: Pharmacokinetics of Afamelanotide in EPP Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinuvel Europe Limited (Industry)
Responsible Party: Sponsor
Organization: Clinuvel Pharmaceuticals Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CUV052
Record Dates: First submitted 2024-04-04; First posted 2024-04-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Erythropoietic Protoporphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide; Drug Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afamelanotide 16 mg implant (Experimental)
  Interventions: Drug: Afamelanotide 16mg implant

INTERVENTIONS:
Drug: Afamelanotide 16mg implant — afamelanotide 16mg implant will be administered to each patient during the study.

SUMMARY:
The purpose of this study is to evaluate the concentration of afamelanotide in serum after the administration of afamelanotide in adolescent and adult EPP patients.

ELIGIBILITY:
Inclusion Criteria:

* EPP patients aged between 12 and 70 years
* BMI between 15 and 30 kg/m2
* >50 kg

Exclusion Criteria:

* Any personal or direct family history of melanoma
* Any significant history of allergy and/or sensitivity to any of the contents of study drug product or lignocaine or other local anaesthetics if used
* Any significant illness during the four weeks before the study screening period
* Any evidence of hepatic or renal impairment

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum Plasma Concentration) | Baseline to Day 7
  Blood samples will be collected for analysis of afamelanotide plasma concentrations and understand what the maximum concentration in plasma is.
AUC(0-t) (area under the curve from administration to last observed concentration at time t) | Baseline to Day 7
  Blood samples will be collected for analysis of afamelanotide plasma concentrations.

SECONDARY OUTCOMES:
AUC(0-∞) (area under the curve extrapolated to infinite time) | Baseline to Day 7

CONTACTS AND LOCATIONS:
Locations (2):
- CLINUVEL Site, Leuven, Belgium
- CLINUVEL Site, Rotterdam, Netherlands